## Study title: Randomized Controlled Trial (RCT) of StriveWeekly for Anxiety and Depression Prevention for College Students During COVID-19

NCT #:NCT04927845

Document date: 06/01/2023

The following "Data analysis" section is an excerpt from a proposal titled "Randomized Controlled Trial of StriveWeekly during COVID-19" that was submitted on 08/14/2020 to Harvard University Foundations of Human Behavior Initiative Proposal.

**Data analysis.** For assessing intervention effects, piecewise LME models will be run in predicting change in outcome scores. Included variables of group, time, group by time interaction, and covariates will be treated as fixed effects, whereas participant intercepts and outcome slopes will be allowed to vary randomly. Between-group and with-group effect sizes (*d*) will be calculated based on estimated marginal means. Moderator and mediator analyses will be selected *post hoc*, based on data completeness. Given the number of exploratory analyses that will be conducted, all significant findings will be tested against Benjamini-Hochberg critical values, on order to control for false discovery rate (i.e., Type I error).